CLINICAL TRIAL: NCT04477226
Title: Pre-Induction Cervical Assessment Using Transvaginal Ultrasound Versus Bishop's Cervical Scoring in Term Pregnancies As Predictors of Successful Induction of Labour
Brief Title: Transvaginal Ultrasound As Predictors of Successful Induction of Labour
Status: Completed | Type: Observational
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: FF-2019-368
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Induction of Labour

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound scan — Transvaginal ultrasound is done to measure the cervical length, as per Fetal Medicine Foundation guidelines

SUMMARY:
To compare the use of transvaginal ultrasound (TVUS) of cervix to the Bishops score prior to induction of labour in term pregnancies, and the ability to predict Caesarean delivery for failure to progress.

DETAILED DESCRIPTION:
The aim of this prospective study is to compare the use of transvaginal ultrasound (TVUS) of cervix to the Bishops score prior to induction of labour in term pregnancies, and the ability to predict Caesarean delivery for failure to progress.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous or multipara
* Singleton live pregnancy
* Gestational age between 37 - 42 weeks
* Cephalic presentation
* Intact membranes
* Reactive cardiotocograph tracing
* Low risk pregnancy

Exclusion Criteria:

* Previous history of uterine surgery
* Low lying placenta, placenta praevia and vaginal bleeding
* Multiple pregnancy
* Preterm Prelabour rupture of membrane/ prelabour rupture of membranes
* Known allergy towards prostaglandins
* Intrauterine fetal death
* Known fetal anomaly
* Estimated fetal weight >3.8kg by scan
* Grandmultiparity (more than 5)
* BMI >40kg/m2
* Diabetes and hypertension on treatment
* Other medical illness on treatment

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — only female pregnant patient
Study Population: All patients who are admitted for induction of labour and fulfils the criteria will be recruited from Patient Admission Centre (PAC), antenatal ward, labour room
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the optimal cutoff points for cervical length measurement as predictor of successful labour induction | before induction of labour
  measurement of cervical length in cm

CONTACTS AND LOCATIONS:
Overall Officials: Kah Teik Chew, Principal Investigator — UKMMC
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No